CLINICAL TRIAL: NCT07349979
Title: Percutaneous Coronary Intervention With Guideline-Directed Medical Therapy Versus Guideline-Directed Medical Therapy Alone for Patients With Ischemic Cardiomyopathy and Reduced Left Ventricular Ejection Fraction: A Randomized, Controlled, Open-Label, Multicenter PCI-GULF Trial
Brief Title: PCI With Guideline-Directed Medical Therapy for HFpEF Patients With Ischemic Cardiomyopathy
Acronym: PCI-GULF
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KY20251223-09; BE2019615 (Other Grant/Funding Number: the Jiangsu Provincial & Nanjing Municipal Clinical Trial Project)
Record Dates: First submitted 2026-01-08; First posted 2026-01-20 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-12

CONDITIONS: Heart Failure With Reduced Ejection Fraction; Coronary Artery Disease
Keywords: HFrEF; PCI; GDMT; MACE
MeSH Terms: conditions — Coronary Artery Disease | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Intervention Model Description: PCI with DES plus GDMT versus GDMT alone
Who Masked: Care Provider, Outcomes Assessor
Masking Description: blinded endpoint adjudication
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- PCI with contemporary DES + GDMT (Experimental): PCI will be performed according to standard techniques. Use of a contemporary, FDA/CE-approved drug-eluting stent is mandatory. Complete revascularization of all angiographically significant lesions (visually estimated stenosis <90% in vessels with RVD ≥2.5 mm and QFR ≤0.80) is encouraged, to be performed either during the index procedure or within a staged procedure within 30 days.
  Post-PCI, dual antiplatelet therapy (DAPT) with aspirin (75-100 mg daily) and a P2Y12 inhibitor (clopidogrel, ticagrelor, or prasugrel per operator choice) will be prescribed for a minimum of 6-12 months, after which single antiplatelet therapy continues indefinitely.
  All subjects receive evidence-based GDMT per guidelines throughout the study.
  Interventions: Procedure: Percutaneous coronary intervention; Drug: Guideline-directed medical therapy
- GDMT only (Active Comparator): The control group will receive GDMT; this is approved treatments for preventing HF that could be utilised as a comparator. All patients will be treated according to local guidelines on standard of care treatment for patients with HFrEF and post PCI, focusing on treatment of HF symptoms (e.g. diuretics) and comorbidities (including treatment for high blood pressure, ischaemic heart disease).
  Interventions: Drug: Guideline-directed medical therapy

INTERVENTIONS:
Procedure: Percutaneous coronary intervention — PCI will be performed according to standard techniques. Use of a contemporary, FDA/CE-approved drug-eluting stent is mandatory.
  Other Names: PCI
  Arms: PCI with contemporary DES + GDMT
Drug: Guideline-directed medical therapy — GDMT optimization follows a structured titration algorithm:
  Week 0: introducing angiotensin-converting enzyme inhibitor (ACEi)/ angiotensin II receptor blocker (ARB) or angiotensin receptor-neprilysin inhibitors (ARNI) and beta-blockers.
  Week 1: adding mineralocorticoid receptor antagonist (MRA) and sodium-glucose cotransporter 2 inhibitors (SGLT2i).
  Adjust every 2-4 weeks to reach target or tolerable dose unless symptomatic hypotension (systolic blood pressure [SBP] < 90 mmHg) or estimated glomerular filtration rate (eGFR) drop > 30 % or serum potassium >5.2 mmol/L.
  Other Names: GDMT

SUMMARY:
To evaluate whether percutaneous coronary intervention (PCI) with contemporary drug-eluting stents (DES) combined with guideline-directed medical therapy (GDMT), compared to GDMT alone, reduces the time to first occurrence of major adverse cardiovascular events (MACE) through 12 months in patients with ischemic cardiomyopathy and a left-ventricular ejection fraction (LVEF) ≤40%. MACE is a composite of cardiovascular [CV] death, spontaneous myocardial infarction (MI), any unplanned revascularization, heart failure (HF)-related rehospitalization, heart transplantation, requirement of device implantation (e.g., valvular treatment, pacemaker, or left ventricular assist device [LVAD]), or requirement of intravenous medications due to worsening heart failure in outpatients.

DETAILED DESCRIPTION:
A prospective, randomized, controlled, open-label, multicenter trial with blinded endpoint adjudication (PROBE design).

A total of 654 patients with LVEF ≤40%, angiographically proven coronary artery disease (CAD) amenable to PCI, and symptomatic heart failure (NYHA Class II-IV) on stable GDMT will be assigned at a 1:1 ratio to:

Experimental Group: PCI with contemporary DES plus GDMT

Control Group: GDMT only

Angiographically proven CAD is defined as a visually estimated diameter stenosis (DS) <90% with a quantitative flow ratio (QFR) ≤0.80 in a major epicardial vessel (reference vessel diameter [RVD] ≥2.5 mm), which is deemed amenable to successful PCI with DES by an interventional cardiologist.

Complete revascularization of all angiographically significant lesions (visually estimated stenosis ≥70% in vessels with RVD ≥2.5 mm) is encouraged, to be performed either during the index procedure or within a staged procedure within 30 days.

Both arms receive optimized GDMT according to current guidelines. Given the nature of the intervention (PCI vs. no PCI), treating physicians and patients cannot be blinded. To minimize bias, a PROBE design is employed with a blinded independent Clinical Events Committee (CEC), blinded core laboratories, and blinded statisticians. The catheterization laboratory team is unblinded but not involved in follow-up decisions or endpoint assessments.

Clinic/telephone follow-up is conducted at 30 days and 3, 6, 9, and 12 months, with annual passive follow-up to 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Both male and female subjects aged ≥18 years at screening.
* Documented LVEF ≤40% assessed by echocardiography, or cardiac magnetic resonance imaging (CMR), or ventriculography within 90 days prior to randomization.
* Symptomatic heart failure (NYHA Functional Class II, III, or ambulatory class IV)
* Angiographically proven CAD with at least one lesion (50~89% stenosis by visual estimate in a major epicardial vessel ≥2.5mm in diameter, or ≥50% left main stenosis, both requiring a QFR≤0.8) considered amenable to PCI with DES by an interventional cardiologist.
* On stable, optimally titrated GDMT for at least 2 weeks prior to randomization, as tolerated. This includes, at a minimum, a beta-blocker and a renin-angiotensin-aldosterone system inhibitor (ACEi/ARB/ARNI) at maximal tolerated doses.
* The subject, or their legal guardian, has a clear understanding of the trial's design and procedures, provides written informed consent, and able to comply with follow-up.

Exclusion Criteria:

* Acute coronary syndrome (ACS) within 30 days requiring urgent/emergent revascularization.
* Non-cardiac life expectancy <1 year at screening (e.g., malignancy, advanced liver disease).
* Coronary anatomy unsuitable for PCI or requiring urgent surgical revascularization (e.g., diameter stenosis ≥90%, diameter stenosis <90% but QFR>0.8, complex multi-vessel disease deemed better suited for coronary artery bypass grafting [CABG] by Heart Team).
* Prior CABG.
* HF due to specific cardiomyopathies, including restrictive/infiltrative cardiomyopathy, active myocarditis, constrictive pericarditis, severe valvular stenosis, or hypertrophic obstructive cardiomyopathy (HOCM).
* Contraindication to GDMT medications, dual antiplatelet therapy, or iodinated contrast.
* Pregnancy, lactation, or women of childbearing potential not using effective contraception. A negative urine pregnancy test is required at each visit for women of childbearing potential.
* Participation in another investigational trial that may interfere with the PCI and GDMT as specified in this protocol.
* Any other circumstances that the investigator deems inappropriate for participation, including but not limited to conditions that may jeopardize patient safety, confound data interpretation, or patients unlikely to comply with study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 654 (Estimated)
Dates: Start 2026-01-30 (Estimated); Primary Completion 2028-01-30 (Estimated); Study Completion 2028-01-30 (Estimated)

PRIMARY OUTCOMES:
Major adverse cardiovascular events | From randomization to the 12-month follow-up period
  MACE is a composite of cardiovascular [CV] death, spontaneous myocardial infarction (MI), any unplanned revascularization, heart failure (HF)-related rehospitalization, heart transplantation, requirement of device implantation (e.g., valvular treatment, pacemaker, or left ventricular assist device [LVAD]), or requirement of intravenous medications due to worsening heart failure in outpatients.

SECONDARY OUTCOMES:
Rate of cardiovascular death plus myocardial infarction and revascularization | From randomization to the 12-month follow-up period
  This endpoint measures the time to first occurrence of any component of the composite of cardiovascular death, myocardial infarction, or unplanned ischemia-driven revascularization.
Rate of cardiovascular death | From randomization to the 12-month follow-up period
  A death that is primarily caused by a cardiovascular event or condition. This includes deaths resulting from acute myocardial infarction, stroke, heart failure, arrhythmias, and other cardiovascular diseases.
Rate of myocardial infarction | From randomization to the 12-month follow-up period
  The diagnosis of an myocardial infarction should be made according to standard clinical practice but is expected to align with the criteria from Fourth Universal Definition of MI, i.e. detection of a rise and/or fall of cardiac biomarkers such as troponin and at least one of the following: typical clinical symptoms, ischaemic ECG findings, imaging evidence of myocardial injury, or detection of an intracoronary thrombus by angiography or autopsy.
Rate of any unplanned revascularization | From randomization to the 12-month follow-up period
  Unplanned revascularization includes all coronary revascularization procedures (PCI/CABG) performed during the study.
Rate of heart failure-related rehospitalization | From randomization to the 12-month follow-up period
  Heart failure readmission is defined as a hospitalization or extended emergency visit due to acute worsening of heart failure, requiring all of the following: a primary HF diagnosis, symptom deterioration, objective evidence of worsening, and intensified HF-specific therapy.
Incidence of device implantation procedure | From randomization to the 12-month follow-up period
  Device implants include valve therapy, pacemakers or left ventricular assistive devices.
Heart transplantation | From randomization to the 12-month follow-up period
  Rate of heart transplantation refers to the frequency at which patients in a study undergo surgical replacement of their native heart with a donor heart.
Rate of worsening heart failure | From randomization to the 12-month follow-up period
  worsening HF including intravenous medications in outpatients.
All-cause mortality | From randomization to the 12-month follow-up period
  All-cause mortality refers to the death of a participant from any cause during the study period.
Change in LVEF | From randomization to the 12-month follow-up period
  Change in LVEF refers to the absolute or relative difference in Left Ventricular Ejection Fraction measured from randomization to the 12-month follow-up period.
Change from baseline in NT-proBNP concentration at 12 months | From randomization to the 12-month follow-up period
  Change in NT-proBNP refers to the absolute or relative difference in NT-proBNP measured from randomization to the 12-month follow-up period.
Total number of (first and recurrent) MACE | From randomization to the 12-month follow-up period
  heart failure and cardiovascular death will be combined to report heart failure-related health status.
Change in Kansas City Cardiomyopathy Questionnaire (KCCQ) | From randomization to the 12-month follow-up period
  The Kansas City Cardiomyopathy Questionnaire Clinical Summary Score (KCCQ-CSS) is a percentage-based health index ranging from 0 to 100, where higher scores indicate better heart failure-related health status.

OTHER OUTCOMES:
Rate of Stroke | From randomization to the 12-month follow-up period
  Rate of stroke refers to the frequency of new, acute cerebrovascular events occurring in a study population.
Rate of Major bleeding | From randomization to the 12-month follow-up period
  Major bleeding is defined as bleeding at BAR 3 grade or above.
Rate of contrast-associated acute kidney injury | Within 48 hours after contrast administration
  Contrast-associated acute kidney injury (CA-AKI), defined according to the PC-AKI criteria as an increase in serum creatinine by ≥26.5 μmol/L or to ≥1.5 times the baseline level within 48 hours after contrast administration.

CONTACTS AND LOCATIONS:
Overall Officials: Shao-Liang Chen, MD, Principal Investigator — Nanjing First Hospital, Nanjing Medical University
Locations (1):
- Nanjing First Hospital, Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No